CLINICAL TRIAL: NCT07169305
Title: Impact of DME on Pulpal and Periodontal Health at Varying Gingival Seat Level in Class II Subgingival Composite Restorations
Brief Title: Impact of DME on Pulpal and Periodontal Health at Varying Gingival Seat Level
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Swathi C
Record Dates: First submitted 2025-05-15; First posted 2025-09-11 (Actual); Last update posted 2025-09-11 (Actual); Status verified 2025-04

CONDITIONS: Deep Margin Elevation; Pulpal and Periodontal Health
Keywords: Deep margin elevation; Pulpal and Periodontal health; Class II Composite restorations

STUDY DESIGN:
Who Masked: Participant
Masking Description: Masking Description
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Class II cavities 2mm to <3mm above the alveolar crest (Experimental): DME is performed in Class II cavities 2mm to <3mm above the alveolar crest and restored with composite.
  Interventions: Procedure: Deep Margin Elevation
- Class II cavities 1mm to <2mm above the alveolar crest (Experimental): DME is performed in Class II cavities 1mm to <2mm above the alveolar crest and restored with composite.
  Interventions: Procedure: Deep Margin Elevation
- Class II cavities ≥3mm above the alveolar crest (Active Comparator): DME is performed in Class II cavities ≥3mm above the alveolar crest and restored with composite.
  Interventions: Procedure: Deep Margin Elevation

INTERVENTIONS:
Procedure: Deep Margin Elevation — The tooth preparation is performed using conventional diamond burs. The extent of caries decides the group into which the participant falls. A precontoured sectional matrix (Palodent) with a properly sized plastic diamond wedge (Bioclear Matrix Systems) is applied and stabilized using a separating ring to ensure closure of deep cervical margins, adaptation of the matrix cervically and attain contact tightness. A 37% phosphoric acid etch gel is used for Selective Enamel Etching technique for 15-20 seconds. Two coats of adhesive are applied to both enamel and dentin using a microbrush and light cured. Flowable bulkfill composite (SDR plus, Dentsply, Sirona) restorative composite is placed using teflon coated hand instruments to perform DME till the level of CEJ and light cured for 20s. Further build up of proximal box is done using packable composite. The restoration is finished using fine grit yellow coded tapered diamond stones. Polishing done by using Composite Polishing kits.

SUMMARY:
The classical idea was to keep the biologic width untouched in order to maintain periodontal health but the newer case reports have given a new dimension to this concept, stating that a limited extension into STA can be used as an alternative for invasive procedures like SCL. The periodontal tissues can still tolerate subgingival margin placement in biologic width when restorations are free of overhangs which are real culprit for providing room for plaque retention and further inflammation. There are no sufficient clinical studies with good sample size to prove the significance of this concept. Hence, we are performing a Non Randomized Controlled trial by placing gingival margins at various levels above the alveolar crest and restoring it with composite and further evaluate the periodontal tissue health, pulpal health, restoration quality and significance of DME.

DETAILED DESCRIPTION:
Rationale: Deep margin Elevation is a technique used in restorative dentistry which helps in dealing with deep Subgingival margins. The placement of gingival seat in relation to crestal bone significantly influences pulpal and periodontal health. Biologic width is essential for maintaining healthy periodontal tissues, but the effect of limited violations needs to be evaluated. Less invasive procedures like DME are preferable alternative to surgical crown lengthening. Aims & Objectives: 1.To evaluate and compare the effect of DME performed in Class II at ≥3mm, 2mm to <3mm, 1mm to <2mm above alveolar crest on pulpal health 2.To evaluate and compare the effect of DME performed in Class II at ≥3mm, 2mm to <3mm, 1mm to <2mm above alveolar crest on gingival health 3.To evaluate and compare the effect of DME performed in Class II at ≥3mm, 2mm to <3mm, 1mm to <2mm above alveolar crest on restoration quality.

Population - Adult patients with class II cavities at ≥3mm, 2mm to <3mm, 1mm to <2mm above the alveolar crest. Intervention - DME performed in Class II cavities at 2mm to <1mm and 1mm to <2mm above the alveolar crest with composite. Comparator- DME performed in Class II cavities at ≥3mm above the alveolar crest with Composite. Outcome- Clinical performance according to USPHS criteria, Periodontal parameters i.e. Probing depth and CAL, Gingival Index and Plaque Index.

ELIGIBILITY:
Inclusion Criteria:

* Patients at least 18 years of age at the time of treatment.

  * Permanent Posterior teeth exhibiting proximal caries lesion extending subgingivally below the cemento-enamel junction (CEJ). The axial extent of the caries should not be more than 75% of the dentin thickness.
  * Sound tooth structure of atleast 1mm should be present from the alveolar crest to the base of the cavity/ gingival seat after cavity preparation.
  * The tooth should either be asymptomatic or have reversible pulpitis as determined by history and pulp sensibility testing. There should be no history of spontaneous or lingering pain
  * Periodontally sound tooth
  * Full mouth plaque score (FMPS): ≤ 15% and Full mouth bleeding score (FMBS): ≤15%

Exclusion Criteria:

* Presence of bone disease (metabolic, endocrine, infectious, tumoral, developmental pathologies)

  * Pregnant or lactating and history of smoking or alcohol abuse
  * Anti inflammatory drug consumption within past 3 days
  * Uncontrolled or poorly controlled diabetes
  * Unstable Life threatening conditions or requiring antibiotic prophylaxis.
  * Presence of detectable plaque and Bleeding on probing on the tooth to be treated
  * Thin gingival biotype, Periodontitis and Gingival recession
  * Class II cavities with gingival margin above the CEJ
  * Previously restored teeth
  * Absence of adjacent tooth or antagonist or Crown in adjacent tooth.
  * H/o Bruxism, Xerostomia
  * Requiring gingivectomy
  * Isolation with rubber dam not possible

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Periodontal Parameters | Baseline to 12 months
  Probing Depth

SECONDARY OUTCOMES:
Periodontal parameters and restoration quality | Baseline to 12 months
  CAL, Plaque Index, Gingival Index. United States Public Health Service (USPHS) criteria for restoration quality

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Mayank Arora, MDS, Principal Investigator — PGIDS, Rohtak
Locations (1):
- PGIDS, Rohtak, Haryana, India